CLINICAL TRIAL: NCT00761020
Title: Analysis of Anti-Plasmodium Falciparum Merozoite Surface Protein 1 Antigen Specific Antibodies in a Human Malaria Challenge Using Mefloquine Prophylaxis to Confirm Assay Sensitivity and Establish Key Antibody Kinetic Parameters
Brief Title: Merozoite Surface Protein 1 Antibody Response in Asymptomatic Human Malaria Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WRAIR 1490; HSRRB Log#A-15136
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Malaria
Keywords: Malaria; Diagnosis; Biomarker
MeSH Terms: conditions — Malaria; Disease | interventions — Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mefloquine (Experimental): Mefloquine 250 mg orally daily x 3 days beginning 2 days prior to challenge and then weekly for 4 weeks post challenge.
  Interventions: Drug: Mefloquine
- Control (Sham Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Drug: Mefloquine — To determine the seroconversion rate (sensitivity) to Plasmodium falciparum Merozoite Surface Protein 1 (Pf MSP-1) antigen by ELISA assay in the infectivity control and mefloquine cohorts as part of a larger project to support the qualification of anti-MSP-1 antigen-specific antibody assays as valid surrogate endpoints for malaria infection.
  Other Names: Lariam
  Arms: Mefloquine
Other: Control — No Intervention
  Arms: Control

SUMMARY:
The main purpose of this trial is to study whether a certain blood test can reliably identify the presence of malaria in people who have been infected with, but who do not have symptoms of malaria.

DETAILED DESCRIPTION:
In this study, two groups of volunteers will be exposed to malaria through the bites of infected mosquitoes. In one group, volunteers will be given several doses of a drug called mefloquine, known to prevent the development of malaria symptoms. The other group will not be treated with any drug that could prevent symptoms or infection. After exposure, both groups will be monitored for a period of approximately 6 months to see if they develop symptoms of malaria. Any subjects who do so will be treated with appropriate medications. Subjects in both groups will have their blood checked regularly during this period for the presence of a certain malaria antibody called Merozoite Surface Protein 1, or Anti-MSP-1 for short, using a special blood test (also known as an assay). At the completion of the study, the results of all assays will be analyzed to determine if this test can be used to diagnose malaria infection in persons without symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant, non-lactating female 18 to 55 years of age (inclusive) at the time of screening
* Written informed consent obtained from the participant before screening procedures
* Free of clinically significant health problems as established by medical history and clinical examination before entering into the study
* Available to participate for duration of study (approximately 6 months, not including screening period)
* If the participant is female, she must be of non-childbearing potential, (i.e., either surgically sterilized or one year post-menopausal) or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or Depo-Provera®) during this study, have a negative pregnancy test at the time of enrollment, and must agree to continue such precautions for at least two months after completion of the malaria challenge if part of the control cohort, or for three months after the final mefloquine dose is taken if part of the mefloquine cohort.
* Prior to entry into this study, participants must score at least 80% correct on a short multiple-choice quiz that assesses their understanding of this study. If they do not score 80% on the initial quiz, the protocol information will be reviewed with them to ensure comprehension and they will have the opportunity to retest (using the same test). Participants who fail the Comprehension Assessment for the second time will not be enrolled.

Exclusion Criteria:

* History of malaria
* Travel to a malarious country within the previous 12 months
* History of participation in a study in which potential exposure to malaria or vaccination against malaria occurred.
* Planned travel to malarious areas during the study period
* History of malaria chemoprophylaxis within 60 days prior to time of study entry
* Recent (defined as any use within 30 days of study entry) or chronic use (defined as more than 14 days of use within 60 days of study entry) of antibiotics with anti-malarial effects (e.g., tetracyclines for dermatologic patients, clindamycin for soft tissue and bone infections, sulfa for recurrent urinary tract infections, etc.)
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of study entry. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Administration of immunoglobulins and/or any blood products within the three months preceding study entry or planned administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Personal medical histories including the following diagnoses: systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, scleroderma, vasculitis, and multiple sclerosis
* Elevated serum creatinine, defined in this study as greater than or equal to 1.7 mg/dL in males and 1.4 mg/dL in females
* Elevated transaminases, defined in this study as greater than twice the upper limit of the normal range (>2 ULN)
* Significant unexplained anemia: hematocrit < 35%
* History of sickle cell disease or sickle cell trait
* Seropositive for hepatitis B surface antigen or hepatitis C antibody
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* History of splenectomy
* Pregnant or lactating female, or female who intends to become pregnant during the study
* Chronic or active neurologic disorders including seizures, excluding a single febrile seizure as a child
* History of a neuropsychiatric disorder (anxiety, depression, psychosis, schizophrenia, PTSD, etc.)
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV (Diagnostic and Statistical Manual of Mental Disorders- 4th edition)
* Chronic or active illicit and/or intravenous drug use
* History of severe anaphylactic reactions to mosquito bites
* History of allergy to mefloquine
* History of intolerance to mefloquine
* History of psoriasis (given its interaction with chloroquine)
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Subjects showing four-fold increase in antibody titer | 1 year
  The focus of the statistical analysis will be to estimate (with 95% confidence limits) the sensitivity of Pf assay in the mefloquine and control arms. Sensitivity will be calculated as the number of subjects in each cohort who develop at least a four-fold increase in antibody titer from baseline (measured positives) divided by the number infected (true positives). The binomial test will used to test the null hypothesis that the sensitivity in the mefloquine arm is at 30% α(= 0.05; one-sided). The control group will serve as a check on the challenge. The study is not powered to statistically test for a difference in sensitivity between mefloquine and control arms. ELISA titer data will be log-transformed for all analyses. For each group, geometric mean anti-MSP-1 antibody titers with 95% confidence intervals will be determined by ELISA and tabulated at each time point which blood samples are taken for serology.

SECONDARY OUTCOMES:
Subjects showing Anti- Pf MSP-1 IgG antibody response | 1 year
  The focus of the statistical analysis will be to characterize the antibody kinetics in subjects over that time, will be presented graphically in whole blood concentration vs. time plots. We will identify individual Cmax, t 1/2, and time to Cmax as well determined point estimates and confidence intervals for the cohorts. We will also estimate the percentage cross-reactivity of the serum in each cohort by measuring the number of subjects who test Pf assay positive divided by the number of subjects Pf infected with in each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: James Moon, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States